CLINICAL TRIAL: NCT03041961
Title: Effects of Aronia Berry (Chokeberry) Extract on Vascular Function in Healthy Men: a 3 Month Randomized Controlled Trial.
Brief Title: Aronia Berry Consumption on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Naturex-Dbs (Industry)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Principal investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Aronia FMD
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy Young Men
Keywords: Vascular function; Endothelial function; (Poly)phenols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Formulation containing inert artificially colored maltodextrin, once daily, in a 1-hard capsule regimen (500 mg)
  Interventions: Dietary Supplement: Placebo
- Aronia full spectrum (Active Comparator): Formulation of an aronia full spectrum ingredient in a 1-hard capsule regimen (500 mg)
  Interventions: Dietary Supplement: Aronia full spectrum
- Aronia extract (Active Comparator): Formulation of an aronia extract ingredient in a 1-hard capsule regimen (500 mg)
  Interventions: Dietary Supplement: Aronia extract

INTERVENTIONS:
Dietary Supplement: Placebo — Identical formulation as the treatment consisting of colored maltodextrin using artificial colors.
  Arms: Placebo
Dietary Supplement: Aronia full spectrum — Powdered whole fruit obtained from aronia berries (Aronia melanocarpa)
  Arms: Aronia full spectrum
Dietary Supplement: Aronia extract — Powdered extract obtained from aronia berries (Aronia melanocarpa)
  Arms: Aronia extract

SUMMARY:
There is an increasing interest in the effects of various food derived polyphenols on vascular function. Arguably the most well-established vascular benefits are attributed to flavanols from cocoa beans and this has been supported by a successful health claim through the European Food Safely Authority in 2012. Berry fruits are another rich source of polyphenols that have vasoactive properties, and there is a growing body of research exploring these effects in various berries (blueberries, cranberries, strawberries) and other fruit products with similar polyphenol composition. A key (poly)phenol in berries and other fruits believed to provide much of the benefit is anthocyanins. When given as an isolated extract, 320 mg anthocyanins have been found to improve blood vessel function both acutely and in response to chronic consumption over 12 weeks.

Aronia berries are a native North American berry with high naturally occurring anthocyanins among other polyphenols. Based on their polyphenol composition, there is growing interest in the potential for Aronia berries to elicit health promoting cardio-metabolic effects. Specifically, Aronia berry extracts, which provide a concentrated source of polyphenols, may improve blood vessel function.

Thus, the primary focus of this project is to evaluate the effects of Aronia berry extracts of differing polyphenol dose on vascular endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 18-45 years old
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Are able to understand the nature of the study
* Able to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Manifest cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral artery disease
* Hypertensive, as defined as SBP superior or equal to 140 mmHg or DBP superior or equal to 90 mmHg
* Obese participants, defined as BMI superior or equal to 30
* Diabetes mellitus and metabolic syndrome
* Acute inflammation
* Terminal renal failure
* Malignancies
* Abnormal heart rhythm (lower or higher than 60-100 bpm)
* Allergies to berries or other significant food allergy.
* Subjects under medication or on vitamin/dietary supplements.
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently in a diet
* Subjects who reported participant in another study within one month before the study start
* Subjects who smoke an irregular amount of cigarettes per day
* Unable to swallow the capsule
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Change form Baseline Endothelial function at 12 weeks

SECONDARY OUTCOMES:
Pulse wave velocity | Baseline and 12 weeks
  Measured by SphygmoCor 0 and 2 hours postconsumption
Blood pressure | Baseline and 12 weeks
  Automatical measurements 0 and 2 hours postconsumption
Blood measurements- Blood lipids | Baseline and 12 weeks
  Cholesterol, HDL, LDL, triglycerides
Blood measurements | Baseline and 12 weeks
  Haematology (White blood cell count, red blood cell count, Haemoglobin, hematocrit, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils, reticulocytes, eosinophils
Blood measurements-Electrolytes | Baseline and 12 weeks
  Urea, Creatinine, uric acid
Blood measurements | Baseline and 12 weeks
  Liver values (bilirubin, lactate dehydrogenase, aspartate aminotransferase, gamma-glutamyltranspeptidase, total protein, albumine, alkaline phosphatase)
Blood measurements -Glucose | Baseline and 12 weeks

OTHER OUTCOMES:
Plasma aronia berry (poly)phenol metabolites | Baseline 0 and 2 hours and 12 weeks 0 and 2 hours
  Measured by liquid chromotography- mass spectrometry (LC/MS) 0 and 2 hours postconsumption
Microbiome analysis | Baseline and 12 weeks
  Stool sample collection (Umnigene gut collection kit)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Life Sciences and Medecine, London, Central London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Istas G, Wood E, Le Sayec M, Rawlings C, Yoon J, Dandavate V, Cera D, Rampelli S, Costabile A, Fromentin E, Rodriguez-Mateos A. Effects of aronia berry (poly)phenols on vascular function and gut microbiota: a double-blind randomized controlled trial in adult men. Am J Clin Nutr. 2019 Aug 1;110(2):316-329. doi: 10.1093/ajcn/nqz075. PMID 31152545